CLINICAL TRIAL: NCT05405231
Title: Connecting National Guard Service Members Through Education in Crisis Line Facilitation Training
Acronym: CONNECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Michigan Army National Guard (Unknown)
Responsible Party: Principal Investigator, Mark A. Ilgen, Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00193639; R49CE003085 (NIH)
Record Dates: First submitted 2022-05-31; First posted 2022-06-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Suicide
Keywords: Training; Crisis Line
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Intervention Model Description: In Phase 1, we will utilize a cluster randomized control trial (RCT) design to recruit from approximately 12 National Guard (NG) units within the Michigan NG. Soldiers from the selected NG units will be approached for study recruitment during their drill weekends. Only units with >25 Soldiers (out of ~110 units in Michigan) will be eligible to be selected for study recruitment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Crisis Line Facilitation (CLF) (Experimental): Crisis Line Facilitation (CLF) is a promising translational strategy designed to increase Military and Veteran's Crisis Line (MVCL) use among NG members during periods of elevated suicidal risk by addressing individual-level barriers.
  Interventions: Behavioral: Crisis Line Facilitation (CLF)
- Passive Implementation (Active Comparator): The PI condition includes an educational resource brochure describing the Military and Veteran's Crisis Line (MVCL), including the phone number for the crisis line, as well as other mental health services available to National Guard members.
  Interventions: Behavioral: Passive Implementation

INTERVENTIONS:
Behavioral: Crisis Line Facilitation (CLF) — Crisis Line Facilitation (CLF) is a promising translational strategy designed to increase MVCL use among NG members during periods of elevated suicidal risk by addressing individual-level barriers.
  Arms: Crisis Line Facilitation (CLF)
Behavioral: Passive Implementation — The PI condition includes an educational resource brochure describing the MVCL, including the phone number for the crisis line, as well as other mental health services available to National Guard members.
  Arms: Passive Implementation

SUMMARY:
National Guard (NG) are affected by suicide at a much higher rate than civilians. The Military and Veterans Crisis Line (MVCL) is not being used as often as we would expect. The purpose of this study is to find out whether a group-based training session will impact awareness and use of the Military and Veterans Crisis Line (MVCL) among members of the National Guard.

ELIGIBILITY:
Inclusion Criteria:

* Michigan Army National Guard member
* Associated with a unit with more than 25 members

Exclusion Criteria:

- Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 538 (Actual)
Dates: Start 2023-02-11 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Utilization of the Military and Veterans Crisis Line (MVCL) | 6 month follow-up
  Utilization is defined by contacting the MVCL via any method (call, text message, or online chat) at least one time following study enrollment. Data will be collected via self-report survey items.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ilgen, PhD, Study Chair — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No